CLINICAL TRIAL: NCT05722015
Title: A Phase 3 Randomized, Open-label Clinical Study to Evaluate the Pharmacokinetics and Safety of Subcutaneous Pembrolizumab Coformulated With Hyaluronidase (MK-3475A) Versus Intravenous Pembrolizumab, Administered With Chemotherapy, in the First-line Treatment of Participants With Metastatic Non-small Cell Lung Cancer
Brief Title: A Study of Subcutaneous (SC) Pembrolizumab Coformulated With Berahyaluronidase Alfa (MK-3475A) vs Intravenous Pembrolizumab in Adult Participants With Metastatic Non-small Cell Lung Cancer (NSCLC) (MK-3475A-D77)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475A-D77; 2022-501506-36-00 (Registry Identifier: EU CT); MK-3475A-D77 (Other: MSD); jRCT2031230049 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); U1111-1280-9384 (Registry Identifier: UTN)
Record Dates: First submitted 2023-01-27; First posted 2023-02-10 (Actual); Results first posted 2025-07-28 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin; Carboplatin; Paclitaxel; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; pembrolizumab; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy (Experimental): Participants with treatment-naïve metastatic NSCLC receive 790 mg of Pembrolizumab Formulated With Berahyaluronidase Alfa via subcutaneous (SC) injection on Day 1 of each 6-week cycle for 18 cycles (up to approximately 108 weeks) in combination with platinum doublet chemotherapy.
  Interventions: Biological: Pembrolizumab Formulated with Berahyaluronidase Alfa; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Filgrastim; Drug: Pegylated filgrastim
- Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy (Active Comparator): Participants with treatment-naïve metastatic NSCLC receive 400 mg pembrolizumab intravenous (IV) infusion in combination with platinum doublet chemotherapy.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel; Biological: Pembrolizumab; Drug: Filgrastim; Drug: Pegylated filgrastim

INTERVENTIONS:
Biological: Pembrolizumab Formulated with Berahyaluronidase Alfa — Pembrolizumab (+) Berahyaluronidase alfa SC will be administered for squamous and nonsquamous NSCLC as per the schedule specified in arm; participants may be eligible for second course.
  Other Names: MK-3475A
  Arms: Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy
Drug: Pemetrexed — Pemetrexed 500 mg/m² by IV Infusion will be administered for nonsquamous NSCLC as per the schedule specified in arm.
  Other Names: Alimta
Drug: Cisplatin — Cisplatin 75 mg/m² by IV Infusion will be administered for nonsquamous and squamous NSCLC as per the schedule specified in arm.
  Other Names: Platinol-AQ
Drug: Carboplatin — Carboplatin AUC 5 mg/mL/min in nonsquamous and AUC 6 mg/mL/min in squamous NSCLC will be administered as per the schedule specified in arm.
Drug: Paclitaxel — Paclitaxel 200 mg/m² by IV Infusion will be administered for squamous NSCLC as per the schedule specified in arm.
  Other Names: Taxol
Drug: Nab-paclitaxel — Nab-paclitaxel 100 mg/m² by IV Infusion will be administered for squamous NSCLC as per the schedule specified in arm.
  Other Names: Albumin-bound paclitaxel
Biological: Pembrolizumab — Pembrolizumab by IV Infusion will be administered for squamous and nonsquamous NSCLC as per the schedule specified in arm; participants may be eligible for second course.
  Other Names: MK-3475, KEYTRUDA
  Arms: Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy
Drug: Filgrastim — Filgrastim will be administered as per the schedule specified for the arm.
Drug: Pegylated filgrastim — Pegylated filgrastim will be administered as per the schedule specified for the arm.

SUMMARY:
This study is to assess the pharmacokinetics (PK) and safety of SC pembrolizumab formulated with berahyaluronidase alfa (MK-3475A) versus (vs) intravenous (IV) pembrolizumab (MK-3475), administered with chemotherapy in first line treatment of adult participants with metastatic non-small cell lung cancer. The primary hypotheses of this study are pembrolizumab formulated with berahyaluronidase alfa subcutaneous (SC) is noninferior to pembrolizumab IV with respect to PK parameters.

ELIGIBILITY:
The key inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has histologically or cytologically confirmed diagnosis of squamous or non-squamous Non-small Cell Lung Cancer (NSCLC)
* Must provide archival tumor tissue sample or newly obtained core, incisional, or excisional biopsy of a tumor lesion not previously irradiated
* Has a life expectancy of at least 3 months

Exclusion Criteria:

* Has a diagnosis of small cell lung cancer or, for mixed tumors, presence of small cell elements
* Has received prior systemic anticancer therapy for metastatic NSCLC
* Has received prior systemic anticancer therapy including investigational agents within 4 weeks before randomization
* Has received prior radiotherapy within 2 weeks of start of study intervention or has radiation-related toxicity requiring corticosteroids
* Has received radiation therapy to the lung (>30 Gray) within 6 months of start of study intervention
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has an active infection requiring systemic therapy
* Has a history of human immunodeficiency virus (HIV) infection
* Has a history of Hepatitis B or C
* Has not adequately recovered from major surgery or has ongoing surgical complications
* Has a history of allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2028-05-22 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (110):
- United States (9):
  - St. Joseph's Hospital and Medical Center-Dignity Health Cancer Institute ( Site 0023), Phoenix, Arizona
  - Clermont Oncology Center ( Site 0018), Clermont, Florida
  - Mid Florida Hematology and Oncology Center ( Site 0010), Orange City, Florida
  - University of Illinois at Chicago-University of Illinois Cancer Center ( Site 0022), Chicago, Illinois
  - Orchard Healthcare Research Inc. ( Site 0011), Skokie, Illinois
  - Franciscan Health Lafayette East ( Site 0020), Lafayette, Indiana
  - Mercy Health-Paducah Cancer Center ( Site 0006), Paducah, Kentucky
  - Hattiesburg Clinic Hematology/Oncology ( Site 0008), Hattiesburg, Mississippi
  - Central Care Cancer Center - Bolivar ( Site 0017), Bolivar, Missouri
- Argentina (7):
  - Hospital Italiano de Buenos Aires-Clinical Oncology ( Site 1005), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 1001), Mar del Plata, Buenos Aires
  - Instituto Argentino de Diagnóstico y Tratamiento (IADT) ( Site 1002), Buenos Aires, Buenos Aires F.D.
  - Instituto Alexander Fleming ( Site 1008), Buenos Aires, Buenos Aires F.D.
  - Clinica Adventista Belgrano-Oncology ( Site 1004), Buenos Aires, Buenos Aires F.D.
  - Sanatorio Parque ( Site 1003), Rosario, Santa Fe Province
  - Hospital Italiano de Córdoba ( Site 1000), Córdoba
- Brazil (5):
  - CRIO - CENTRO REGIONAL INTEGRADO DE ONCOLOGIA-Pesquisa Clínica ( Site 1102), Fortaleza, Ceará
  - Hospital de Cancer de Pernambuco ( Site 1107), Recife, Pernambuco
  - Hospital Nossa Senhora da Conceição-Centro Integrado de Pesquisa em Oncologia ( Site 1100), Porto Alegre, Rio Grande do Sul
  - Instituto Joinvilense de Hematologia e Oncologia ( Site 1101), Joinville, Santa Catarina
  - A. C. Camargo Cancer Center ( Site 1106), São Paulo
- Chile (7):
  - IC La Serena Research ( Site 1207), La Serena, Coquimbo Region
  - Oncocentro Valdivia ( Site 1201), Valdivia, Los Ríos Region
  - FALP-UIDO ( Site 1203), Santiago, Region M. de Santiago
  - Oncovida ( Site 1209), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile-Hemato-Oncology ( Site 1210), Santiago, Region M. de Santiago
  - Instituto Nacional del Cancer-CR Investigación ( Site 1211), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 1202), Santiago, Region M. de Santiago
- China (17):
  - Anhui Provincial Hospital-Cancer Chemotherapy Department ( Site 4503), Hefei, Anhui
  - Beijing Cancer hospital-intrathoratic deparmtment II ( Site 4510), Beijing, Beijing Municipality
  - Beijing Peking Union Medical College Hospital-pneumology department ( Site 4501), Beijing, Beijing Municipality
  - Beijing Chest Hospital,Capital Medical University ( Site 4511), Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital ( Site 4516), Wanzhou, Chongqing Municipality
  - Fujian Provincial Cancer Hospital ( Site 4517), Fuzhou, Fujian
  - Southern Medical University Nanfang Hospital-Depatrment of Respiratory and Critical Care Medicine ( Site 4519), Guangzhou, Guangdong
  - Jiangmen Center Hospital ( Site 4509), Jiangmen, Guangdong
  - ShenZhen People's Hospital ( Site 4504), Shenzhen, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology-Medical Oncology ( Site 4502), Wuhan, Hubei
  - The First Affiliated Hospital of Nanchang University-Respiratory Medicine Department ( Site 4515), Nanchang, Jiangxi
  - The First Affiliated Hospital of Xi'an Jiaotong University ( Site 4520), Xi'an, Shaanxi
  - Fudan University Shanghai Cancer Center-Oncology ( Site 4512), Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital ( Site 4521), Taiyuan, Shanxi
  - Tianjin Chest Hospital ( Site 4518), Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University-Respiratory Department ( Site 4514), Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province ( Site 4508), Linhai, Zhejiang
- France (3):
  - Centre Hospitalier de Cornouaille Quimper - Concarneau ( Site 2600), Quimper, Finistere
  - Centre Hospitalier Régional Universitaire de Tours - Hôpital Bretonneau ( Site 2602), Tours, Indre-et-Loire
  - Hopitaux Universitaires Paris Centre-Hopital Cochin ( Site 2603), Paris
- Guatemala (4):
  - MEDI-K ( Site 1403), Guatemala City
  - Private Practice- Dr. Rixci Augusto Lenin Ramírez ( Site 1404), Guatemala City
  - Centro Regional de Sub Especialidades Médicas SA ( Site 1401), Quetzaltenango
  - Centro Medico Integral De Cancerología (CEMIC) ( Site 1400), Quetzaltenango
- Hungary (5):
  - Bacs-Kiskun Megyei Korhaz-Onkoradiologiai Kozpont ( Site 2102), Kecskemét, Bács-Kiskun county
  - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház-Onkologiai Kozpont ( Site 2103), Szolnok, Jász-Nagykun-Szolnok
  - Reformatus Pulmonologiai Centrum ( Site 2105), Törökbálint, Pest County
  - Semmelweis Egyetem-Pulmonológiai Klinika ( Site 2104), Budapest
  - Országos Korányi Pulmonológiai Intézet-VI. Tüdöbelosztály és Bronchológia ( Site 2100), Budapest
- Japan (18):
  - Fujita Health University Hospital ( Site 4406), Toyoake, Aichi-ken
  - Kurume University Hospital ( Site 4412), Kurume, Fukuoka
  - Gunma Prefectural Cancer Center ( Site 4416), Ōta, Gunma
  - National Hospital Organization Hokkaido Cancer Center ( Site 4415), Sapporo, Hokkaido
  - Kanagawa Cardiovascular and Respiratory Center ( Site 4404), Yokohama, Kanagawa
  - Miyagi Cancer Center ( Site 4401), Natori-shi, Miyagi
  - Sendai Kousei Hospital ( Site 4400), Sendai, Miyagi
  - Kurashiki Central Hospital ( Site 4409), Kurashiki, Okayama-ken
  - Kansai Medical University Hospital ( Site 4408), Hirakata, Osaka
  - Osaka Medical and Pharmaceutical University Hospital ( Site 4414), Takatsuki, Osaka
  - Saitama Prefectural Cancer Center ( Site 4402), Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center ( Site 4405), Sunto-gun,, Shizuoka
  - Tochigi Cancer Center ( Site 4417), Utsunomiya, Tochigi
  - Juntendo University Hospital ( Site 4413), Bunkyo-ku, Tokyo
  - National Hospital Organization Kyushu Medical Center ( Site 4411), Fukuoka
  - National Hospital Organization Kyushu Cancer Center ( Site 4410), Fukuoka
  - Osaka International Cancer Institute ( Site 4407), Osaka
  - Nippon Medical School Hospital ( Site 4403), Tokyo
- Poland (3):
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworow Pluca i Klatki Pier ( Site 2800), Warsaw, Masovian Voivodeship
  - Warmińsko - Mazurskie Centrum Chorób Płuc w Olsztynie-Oddzial Onkologii z Pododdzialem Chemioterapii ( Site 2802), Olsztyn, Warmian-Masurian Voivodeship
  - Szpital Wojewódzki im. Mikoaja Kopernika w Koszalinie-Oddzial Dzienny Chemioterapii ( Site 2801), Koszalin, West Pomeranian Voivodeship
- Romania (4):
  - SC Radiotherapy Center Cluj SRL-Oncologie Medicala ( Site 2303), Florești, Cluj
  - Centrul de Oncologie Sfantul Nectarie-Medical ( Site 2301), Craiova, Dolj
  - Cabinet Medical Oncomed ( Site 2305), Timișoara, Timiș County
  - Institutul Oncologic-Oncologie Medicala ( Site 2302), Cluj-Napoca
- South Africa (6):
  - CANCERCARE LANGENHOVEN DRIVE ONCOLOGY CENTRE ( Site 2903), Port Elizabeth, Eastern Cape
  - Medical Oncology Centre of Rosebank ( Site 2907), Johannesburg, Gauteng
  - Steve Biko Academic Hospital-Medical Oncology ( Site 2904), Pretoria, Gauteng
  - Sandton Oncology Medical Group (Pty) Ltd-Research ( Site 2900), Sandton, Gauteng
  - The Oncology Centre ( Site 2901), Durban, KwaZulu-Natal
  - Cape Town Oncology Trials ( Site 2902), Cape Town, Western Cape
- Spain (4):
  - CHUS - Hospital Clinico Universitario-Servicio de Oncologia ( Site 2404), Santiago de Compostela, La Coruna
  - HOSPITAL GENERAL UNIVERSITARIO GREGORIO MARAÑON-ONCOLOGY ( Site 2401), Madrid, Madrid, Comunidad de
  - Hospital Universitari Vall d'Hebron-Oncology ( Site 2400), Barcelona
  - Hospital Universitario Juan Ramon Jimenez-Oncología Medica ( Site 2402), Huelva
- Taiwan (7):
  - National Taiwan University Cancer Center (NTUCC) ( Site 4205), Taipei City, Taipei
  - Changhua Christian Hospital ( Site 4203), Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital ( Site 4207), Kaohsiung City
  - E-Da hospital ( Site 4208), Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung ( Site 4200), Kaohsiung City
  - National Cheng Kung University Hospital ( Site 4202), Tainan
  - National Taiwan University Hospital-Oncology ( Site 4204), Taipei
- Thailand (4):
  - Chulalongkorn University ( Site 4301), Bangkok, Bangkok
  - Division of Medical Oncology, Siriraj H ( Site 4303), Bangkok, Bangkok
  - Songklanagarind hospital ( Site 4302), Songkhla, Changwat Songkhla
  - Maharaj Nakorn Chiang Mai Hospital ( Site 4300), Chiang Mai
- Turkey (Türkiye) (7):
  - Gulhane Egitim Arastirma Hastanesi-Oncology ( Site 2504), Ankara
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 2506), Ankara
  - Ankara City Hospital-Medical Oncology ( Site 2501), Ankara
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 2502), Istanbul
  - I.E.U. Medical Point Hastanesi-Oncology ( Site 2507), Izmir
  - Memorial Kayseri Hastanesi ( Site 2500), Kayseri
  - İnönü Üniversitesi Turgut Özal Tıp Merkezi-medical oncology depertmant ( Site 2503), Malatya

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Felip E, Rojas CI, Schenker M, Kowalski DM, Casarini IA, Csoszi T, Sendur MAN, Martins J, Calles Blanco A, Wang CC, Wang M, Ramirez Fallas RAL, Yoshioka H, Nair S, Song X, Deng X, Lala M, Eiras R, Takahashi T. Subcutaneous versus intravenous pembrolizumab, in combination with chemotherapy, for treatment of metastatic non-small-cell lung cancer: the phase III 3475A-D77 trial. Ann Oncol. 2025 Jul;36(7):775-785. doi: 10.1016/j.annonc.2025.03.012. Epub 2025 Mar 27. PMID 40157574
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26349&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All randomized participants.
Period: Overall Study
Arm/Group | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy
Started | 251 | 126
Completed | 0 | 0
Not Completed | 251 | 126
Not completed — Death | 57 | 37
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Participants Ongoing | 188 | 88

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy | Total
Number analyzed (Participants) | 251 | 126 | 377
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (9.6) | 64.8 (8.5) | 64.8 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 40 | 109
  Male | 182 | 86 | 268
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 74 | 41 | 115
  Not Hispanic or Latino | 177 | 85 | 262
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 4 | 6
  Asian | 74 | 36 | 110
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 158 | 78 | 236
  More than one race | 12 | 3 | 15
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cycle 1: Area Under the Curve From Time 0 to 6 Weeks (AUC0-6 Weeks) of Pembrolizumab After the First Dose
Description: AUC0-6 weeks was defined as a measure of pembrolizumab exposure that was calculated as the product of serum drug concentration and time from zero to 6 weeks. Blood samples were collected at pre-specified timepoints to determine AUC0-6 weeks. Per protocol, geometric mean AUC0-6 weeks value of pembrolizumab after the first dose of pembrolizumab formulated with berahyaluronidase alfa in arm 1 and after first dose of pembrolizumab in arm 2 was presented.
Time Frame: Cycle 1: Arm 1: Day 1: Predose and Days 2, 3, 4, 5, 6, 7, 10, 15, 29, and 42 postdose; Arm 2: Day 1: Predose and at the end of infusion, Days 4, 15, 29, and 42 postdose (cycle length = 42 days)
Population: All randomized participants who received a dose in Cycle 1 with at least 1 valid postdose pharmacokinetic (PK) sample available in Cycle 1 and for whom a model-based assessment of AUC0-6 weeks could be made.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg·day/mL
Arm/Group | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy
Number analyzed (Participants) | 245 | 126
μg·day/mL | 1633.24 (40.41) | 1437.58 (26.23)
Statistical Analysis 1: Comparison: Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy vs Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy; Test type: Non-Inferiority — Non-inferiority margin is 0.8; p < 0.00001, Welch's t test; One-sided p-value was calculated using the Welch's t test; Geometric Mean Ratio (GMR) = 1.14, 96% CI 2-sided [1.06 to 1.22] — GMR was calculated as the ratio of geometric mean (GM) of Cycle 1 AUC0-6 weeks in Arm 1 to that of Arm 2. The associated 96% confidence interval (CI) were calculated using Welch's t test

2. Primary Outcome: Cycle 3: Trough Serum Concentration (Ctrough) of Pembrolizumab at Steady State
Description: Ctrough was defined as the lowest serum concentration of pembrolizumab reached at steady state. Blood samples were collected at pre-specified timepoints for the determination of Ctrough. Per protocol, geometric mean Ctrough value of pembrolizumab at steady state of pembrolizumab formulated with berahyaluronidase alfa in arm 1 and of pembrolizumab in arm 2 was presented.
Time Frame: Cycle 3: Arm 1: Day 1: Predose and Days 4, 10, and 42 postdose; Arm 2: Day 1: Predose and at the end of infusion, Days 4 and 42 postdose (cycle length = 42 days)
Population: All randomized participants who received a dose in Cycle 1 and Cycle 3 with at least 1 valid postdose PK sample available in Cycle 1 through Cycle 3 and for whom a model-based assessment of Ctrough could be made.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy
Number analyzed (Participants) | 202 | 101
μg/mL | 39.23 (43.29) | 23.49 (44.23)
Statistical Analysis 1: Comparison: Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy vs Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy; Test type: Non-Inferiority — Non-inferiority margin is 0.8; p < 0.00001, Welch's t test; One sided p-value was calculated using Welch's t test; GMR = 1.67, 94% CI 2-sided [1.52 to 1.84] — GMR was calculated as the ratio of GM of Cycle 3 Ctrough in Arm 1 to that of Arm 2. The associated 94% CI were calculated using Welch's t test

3. Secondary Outcome: Cycle 1: Maximum Serum Concentration (Cmax) of Pembrolizumab After the First Dose
Description: Cmax was defined as the maximum serum concentration of pembrolizumab reached after first dose. Blood samples were collected at pre-specified timepoints for the determination of Cmax. Per protocol, geometric mean Cmax value of pembrolizumab after the first dose of pembrolizumab formulated with berahyaluronidase alfa in arm 1 and after first dose of pembrolizumab in arm 2 was presented.
Time Frame: as for outcome 1
Population: All randomized participants who received a dose in Cycle 1 with at least 1 valid postdose PK sample available in Cycle 1 and for whom a model-based assessment of Cmax could be made.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy
Number analyzed (Participants) | 245 | 126
μg/mL | 64.88 (44) | 129.7 (20.8)

4. Secondary Outcome: Cycle 1: Trough Serum Concentration (Ctrough) of Pembrolizumab After the First Dose
Description: Ctrough was defined as the lowest serum concentration of pembrolizumab reached after first dose. Blood samples were collected at pre-specified timepoints for the determination of Ctrough. Per protocol, geometric mean Ctrough value of pembrolizumab after the first dose of pembrolizumab formulated with berahyaluronidase alfa in arm 1 and after first dose of pembrolizumab in arm 2 was presented.
Time Frame: as for outcome 1
Population: All randomized participants who received a dose in Cycle 1 with at least 1 valid postdose PK sample available in Cycle 1 and for whom a model-based assessment of Ctrough could be made.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy
Number analyzed (Participants) | 245 | 126
μg/mL | 19.36 (52.2) | 12.26 (50.8)

5. Secondary Outcome: Cycle 3: Area Under the Curve From Time 0 to 6 Weeks (AUC0-6 Weeks) of Pembrolizumab at Steady State
Description: AUC0-6 weeks was defined as a measure of pembrolizumab exposure that was calculated as the product of serum drug concentration and time from zero to 6 weeks. Blood samples were collected at pre-specified timepoints to determine AUC0-6 weeks. Per protocol, geometric mean AUC0-6 weeks value of pembrolizumab at steady state of pembrolizumab formulated with berahyaluronidase alfa in arm 1 and pembrolizumab in arm 2 was presented.
Time Frame: as for outcome 2
Population: All randomized participants who received a dose in Cycle 1 and Cycle 3 with at least 1 valid postdose PK sample available in Cycle 1 through Cycle 3 and for whom a model-based assessment of AUC0-6 weeks could be made.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg·day/mL
Arm/Group | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy
Number analyzed (Participants) | 202 | 101
μg·day/mL | 2798 (35.5) | 2122 (27.8)

6. Secondary Outcome: Cycle 3: Maximum Serum Concentration (Cmax) of Pembrolizumab at Steady State
Description: Cmax was defined as the maximum serum concentration of pembrolizumab reached at steady state. Blood samples were collected at pre-specified timepoints to determine Cmax. Per protocol, geometric mean Cmax value of pembrolizumab at steady state of pembrolizumab formulated with berahyaluronidase alfa in arm 1 and pembrolizumab in arm 2 was presented.
Time Frame: as for outcome 2
Population: All randomized participants who received a dose in Cycle 1 and Cycle 3 with at least 1 valid postdose PK sample available in Cycle 1 through Cycle 3 and for whom a model-based assessment of Cmax could be made.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy
Number analyzed (Participants) | 202 | 101
μg/mL | 98.96 (36.8) | 148 (21.6)

7. Secondary Outcome: Number of Participants Who Test Positive for Anti-Drug Antibodies (ADAs) for Pembrolizumab
Description: Blood samples were collected at designated time points for the determination of the presence or absence of anti-pembrolizumab antibodies. Per protocol, the number of participants who developed anti pembrolizumab antibodies were reported.
Time Frame: Predose and Postdose on Day 1 of Cycles 1 through 18 (up to approximately 28 months). Each cycle is 6 weeks.
Reporting Status: Not Posted

8. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experienced CR or PR as assessed by Blinded Independent Central Review (BICR) were presented.
Time Frame: Up to approximately 28 months
Reporting Status: Not Posted

9. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by RECIST 1.1. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR were presented.
Time Frame: Up to approximately 28 months
Reporting Status: Not Posted

10. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: Up to approximately 28 months
Reporting Status: Not Posted

11. Secondary Outcome: Duration of Response (DOR)
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until PD or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR were presented.
Time Frame: Up to approximately 28 months
Reporting Status: Not Posted

12. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experienced at least one AE were reported .
Time Frame: Up to approximately 28 months
Reporting Status: Not Posted

13. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported for Arms 1 and 2.
Time Frame: Up to approximately 28 months
Reporting Status: Not Posted

14. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment (EORTC) Quality of Life Questionnaire-Core30 (QLQ-C30) Combined Global Health Status/Quality of Life (Items 29 & 30) Scale Combined Score
Description: EORTC QLQ-C30 is a questionnaire to assess the overall quality of life (QoL) of cancer patients. Participant responses to questions regarding Global Health Status (GHS; "How would you rate your overall health during the past week?") and QoL ("How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1= Very poor to 7=Excellent). The combined score of GHS (Item 29) and QoL (Item 30) is computed by averaging the raw scores of the 2 items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. Per protocol, the change from baseline in GHS and QoL combined score was presented.
Time Frame: Baseline and Week 24
Reporting Status: Not Posted

15. Secondary Outcome: Change From Baseline in Physical Functioning (EORTC-QLQ-C30 Items 1-5) Score
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to 5 questions about their physical functioning (Items 1 to 5) are scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score of items 1 to 5 was computed by averaging the raw scores of the 5 items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. Per protocol, the change from baseline in EORTC QLQ-C30 physical functioning (Items 1-5) combined score was presented.
Time Frame: Baseline and Week 24
Reporting Status: Not Posted

16. Secondary Outcome: Change From Baseline in the European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire C30 (QLQ-C30) Role Functioning Score-Items 6 and 7
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to the questions "Were you limited in doing either your work or other daily activities during the past week?" and "Were you limited in pursuing your hobbies or other leisure time activities during the past week?" will be scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score of items 1 to 5 was computed by averaging the raw scores of the 2 items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. Higher scores indicate a better level of role functioning. Change from baseline in the EORTC QLQ-C30 role functioning (Items 6-7) combined score was presented.
Time Frame: Baseline and Week 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to approximately 16 months
Description: All-Cause Mortality includes all randomized participants. Serious and Other adverse events (AEs) include all randomized participants who received ≥1 dose of study drug. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs. Data are reported by treatment received.
Arm/Group | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy
All-Cause Mortality (participants affected / at risk) | 61/251 | 37/126
Serious Adverse Events (participants affected / at risk) | 98/251 | 51/126
Other Adverse Events (participants affected / at risk) | 236/251 | 123/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy (N=251) | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy (N=126)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 6 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 10 (10) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 7 (8) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (11) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 2 (2)
Immune-mediated hypophysitis (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (2)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 4 (4) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Myiasis (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 25 (26) | 13 (13)
Pneumonia bacterial (Infections and infestations) | 3 (3) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 2 (2)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 1 (1)
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripheral nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arterial thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Pembrolizumab Formulated With Berahyaluronidase Alfa + Platinum Doublet Chemotherapy (N=251) | Arm 2: Pembrolizumab + Platinum Doublet Chemotherapy (N=126)
Anaemia (Blood and lymphatic system disorders) | 146 (220) | 85 (111)
Leukopenia (Blood and lymphatic system disorders) | 74 (192) | 33 (95)
Neutropenia (Blood and lymphatic system disorders) | 105 (230) | 40 (91)
Thrombocytopenia (Blood and lymphatic system disorders) | 71 (126) | 35 (62)
Hyperthyroidism (Endocrine disorders) | 20 (20) | 6 (6)
Hypothyroidism (Endocrine disorders) | 35 (35) | 15 (15)
Constipation (Gastrointestinal disorders) | 35 (41) | 23 (28)
Diarrhoea (Gastrointestinal disorders) | 36 (45) | 17 (22)
Nausea (Gastrointestinal disorders) | 63 (83) | 30 (38)
Vomiting (Gastrointestinal disorders) | 23 (30) | 8 (9)
Asthenia (General disorders) | 24 (24) | 16 (18)
Chest pain (General disorders) | 14 (14) | 2 (2)
Fatigue (General disorders) | 40 (47) | 17 (19)
Oedema peripheral (General disorders) | 15 (15) | 8 (8)
Pyrexia (General disorders) | 19 (20) | 13 (17)
Upper respiratory tract infection (Infections and infestations) | 16 (17) | 8 (9)
Alanine aminotransferase increased (Investigations) | 44 (67) | 18 (28)
Aspartate aminotransferase increased (Investigations) | 47 (69) | 18 (29)
Blood alkaline phosphatase increased (Investigations) | 18 (24) | 13 (19)
Blood creatinine increased (Investigations) | 18 (19) | 12 (15)
Blood lactate dehydrogenase increased (Investigations) | 16 (24) | 10 (13)
Gamma-glutamyltransferase increased (Investigations) | 17 (22) | 8 (11)
Lymphocyte count decreased (Investigations) | 25 (47) | 9 (10)
Weight decreased (Investigations) | 22 (28) | 10 (10)
Decreased appetite (Metabolism and nutrition disorders) | 28 (32) | 27 (30)
Hyperglycaemia (Metabolism and nutrition disorders) | 28 (45) | 13 (20)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 30 (37) | 16 (21)
Hypocalcaemia (Metabolism and nutrition disorders) | 13 (13) | 5 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 21 (25) | 11 (14)
Hyponatraemia (Metabolism and nutrition disorders) | 17 (21) | 13 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (21) | 15 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 12 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (11) | 7 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (9) | 8 (8)
Dizziness (Nervous system disorders) | 15 (15) | 7 (8)
Neuropathy peripheral (Nervous system disorders) | 12 (13) | 7 (7)
Insomnia (Psychiatric disorders) | 13 (13) | 10 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (21) | 11 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 9 (12)
Alopecia (Skin and subcutaneous tissue disorders) | 22 (22) | 13 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 29 (36) | 16 (19)
Rash (Skin and subcutaneous tissue disorders) | 24 (25) | 12 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study may be published or presented at scientific meetings. The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. Any information identified by the Sponsor as confidential must be deleted prior to submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/15/NCT05722015/Prot_SAP_000.pdf